CLINICAL TRIAL: NCT03098823
Title: A Randomized, Double-Blind, Active Comparator-Controlled, Crossover Study to Assess the Capacity of RAYOS® Compared to Immediate-Release Prednisone to Improve Fatigue and Control Morning Symptoms in Subjects With Systemic Lupus Erythematosus
Brief Title: A Crossover Study to Compare RAYOS to IR Prednisone to Improve Fatigue and Morning Symptoms for SLE
Acronym: RIFLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ampel BioSolutions, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMP-002
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Lupus Erythematosus, Systemic; Lupus Erythematosus; Fatigue
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Fatigue | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RAYOS® (Experimental)
  Interventions: Drug: RAYOS
- IR prednisone (Active Comparator)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: RAYOS — FDA approved RAYOS for indication of fatigue in Lupus.
  Arms: RAYOS®
Drug: Prednisone — FDA approved corticosteroid frequently used for SLE.
  Arms: IR prednisone

SUMMARY:
To compare the effect of RAYOS® versus immediate-release (IR) prednisone on fatigue as measured by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent agreeing to all study procedures, before any study-specific procedures are done.
2. Males or non-pregnant females, aged 18 years or older
3. Diagnosis of SLE by either the American College of Rheumatology (ACR) or Systemic Lupus International Collaborating Clinics Classification (SLICC) criteria
4. Fatigue measured by FACIT-F ≤30.
5. On a stable regimen of IR prednisone (5 to 15 mg/day) for a period of at least 30 days prior to Screening, expected to remain stable for the next 6 months.
6. On a stable SLE treatment regimen for a period of at least 30 days prior to Screening, and expected to remain stable for the next 6 months. Any of the following medications are permitted if stable for at least 30 days prior to Screening and expected to remain stable for the next 6 months:

   * Hydroxychloroquine or equivalent anti-malarial
   * Other immunosuppressive or immunomodulatory agents including methotrexate, azathioprine, leflunomide, mycophenolate (including mycophenolate sodium or mycophenylate mofetil at no more than 2 grams/day), belimumab, cyclophosphamide, calcineurin inhibitors (e.g. tacrolimus, cyclosporine)
7. Entry of daily ePRO data on 11 of 14 days during the baseline period, and completion of at least 6 out of the 8 weekly ePRO questionnaires during the baseline period
8. Willing and able to perform and comply with all study procedures, including taking pills daily as prescribed, completing the ePROs on the smart phone, wearing the smart watch day and night, bringing the smartphone on all activities away from home (e.g., walks, errands, visiting, shopping, traveling), keeping the smartphone and smartwatch charged daily, carefully using the smartphone and smartwatch as clinical tools and keeping them secure from others, and attending monthly clinic visits as scheduled
9. Females of childbearing potential must be currently using a highly effective method of contraception that may include, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with vasectomized partner, hysterectomy, bilateral tubal ligation, licensed hormonal methods, intrauterine device, or use of a spermicide combined with a barrier method (e.g., condom, diaphragm) for 30 days before and 90 days after receiving the study drug

Exclusion Criteria:

1. Previously taken any of the following medications:

   * RAYOS®
   * Rituximab within 6 months prior to Screening
   * Any investigational therapy within 3 months or 5 half-lives of the agent prior to Screening
2. History of noncompliance with taking pills as prescribed.
3. Rapidly progressive neurologic disease
4. Rapidly progressive renal disease (defined by proteinuria >6 g/24 hours or equivalent using spot urine protein to creatinine ratio, or serum creatinine >2.5 mg/dL)
5. Diagnosis of fibromyalgia
6. Any of the following clinical laboratory abnormalities:

   * Hemoglobin <8.0 mg/dL
   * Platelet count <50,000/mm3
   * White blood count (WBC) ≤ 2000/mm3; may be 1999-1000/mm3 if stable and related to SLE
   * Absolute neutrophil count (ANC) ≤1000/mm3; may be 500-999/mm3 if stable and related to SLE
   * Aspartate transaminase (AST) or alanine transaminase (ALT) ≥3× upper limit of normal (ULN) unless related to SLE
   * Calculated creatinine clearance ≤25 mL/min per 1.73 m2 (by Cockcroft-Gault equation)
7. Grade 3 or greater laboratory abnormality based on the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE; Appendix 3) except for the following that are allowed:

   * Activated partial thromboplastin time (PTT) > >2.5× ULN due to lupus anticoagulant and not related to liver disease or anti-coagulant therapy
   * Hypoalbuminemia <2 g/dL due to chronic lupus nephritis, and not related to liver disease
   * Gamma glutamyl transferase (GGT) <20× ULN due to lupus hepatitis, and not related to alcoholic liver disease, uncontrolled diabetes, or viral hepatitis. If present, any abnormalities in the ALT and/or AST must be ≤5× ULN
8. Pregnant or nursing, or females not using effective contraception
9. Current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 1 year prior to Screening
10. Clinical evidence of significant unstable or uncontrolled acute or chronic diseases not caused by SLE (e.g., diabetes, cardiovascular, pulmonary, hematologic, gastrointestinal, neurological, or infectious) which, in the opinion of the Investigator, could confound the results of the study or put the subject at undue risk

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Fatigue | 3 months
  Fatigue as measured in FACIT-F by patient

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - The Regents of the University of California, Los Angeles, Los Angeles, California
  - University of California-Irvine, Orange, California
  - Stanford University, Palo Alto, California
  - The Regents of the University of California, San Diego, San Diego, California
  - University of California-San Francisco, San Francisco, California
  - Yale School of Medicine, New Haven, Connecticut
  - University of Florida College of Medicine, Gainesville, Florida
  - Miller School of Medicine at the University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMASS Memorial Medical Center-Memorial Campus, Worcester, Massachusetts
  - The Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The MetroHealth System, Cleveland, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Hershey Medical Center, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No